CLINICAL TRIAL: NCT04569500
Title: FRENCH THERAPEUTIC EDUCATION PROGRAM AIMING TO IMPROVE LARYNGECTOMIZED PATIENTS' AND THEIR FAMILY CAREGIVER'S QUALITY OF LIFE
Acronym: PETAL2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-133
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Patients With Total Laryngectomy and Their Close Relatives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PETAL program (Experimental): Patients with total laryngectomy and their close relatives, benefiting from the therapeutic education program PETAL
  Interventions: Other: PETAL program
- Usual care (No Intervention): Patients with total laryngectomy and their close relatives, benefiting from the usual care

INTERVENTIONS:
Other: PETAL program — patients and their close relations will benefit from the therapeutic education program PETAL in order to accompany them throughout their experience of laryngectomy and to reduce its impact on social and professional aspects of life.
  Arms: PETAL program

SUMMARY:
The therapeutic education of patients and their close relations is, as yet, poorly developed in France in the field of oncology (Pérol2007), in particular for cancers of the upper aerodigestive tract (Allison2010). In the case of pharyngeal and laryngeal cancer, total laryngectomy associated with radiotherapy remains a reference treatment for advanced stage cancers. This mutilating surgical procedure has a major impact on the patient's life, due to its physical and functional sequelae: phonatory (loss of physiological voice), feeding, olfactory and aesthetic (tracheostomy). Its psychosocial consequences are also important, owing to the biographical disruption and the identity-related metamorphoses associated with illness and its treatment, which alter the quality of life not only of patients, but also of their close relations. Indeed, transformation is not only at individual level, it also impacts the life of close relations, in particular spouses, who share the day-to-day lives of patients (Babin 2010). Currently, care for laryngectomized patients consist essentially in informing and educating them on certain technical procedures (cannula replacement, mucosity aspiration, tracheostomy or phonatory implant cleaning) during hospital admission. Such education may be formalized and dispensed within the context of a therapeutic education program.

The issue of this study will be to determine what therapeutic education program we should offer patients and their close relations in order to accompany them throughout their experience of laryngectomy and to reduce its impact on social and professional aspects of life.

ELIGIBILITY:
Patient inclusion criteria

* Patients over 18 having been treated by total laryngectomy for cancer of the larynx, pharynx or cervical esophagus.
* Patients accepting to participate in the study (informed consent form explained and signed).
* Patient having not been undergone a PTE
* Person affiliated with an appropriate social security system.

Close relation inclusion criteria

* Person over 18 designated as being a close relation by the laryngectomized patient (confidential person, spouse, parent, natural support person or any person whose quality of life may be impacted by the patient's laryngectomy).
* Close relation accepting to participate in the study (informed consent form explained and signed).
* Person authorized by the patient to be contacted by the investigator, in order to propose his/her participation in the research study.
* Person affiliated with an appropriate social security system.

Patient exclusion criteria - Physical, psychical, psychiatric or cognitive incapacity to answer to questions or participate in interviews/sessions.

Close relation exclusion criteria

- Physical, psychical, psychiatric or cognitive incapacity to answer to questions or participate in interviews/sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life score (PSS-HN scale) of patients with total laryngectomy | 12 months
  Difference in gain observed at six months in the mean quality of life score (PSS-HN scale) of patients with total laryngectomy and their close relatives, having benefited from the PTE program and those having benefited from usual care.

SECONDARY OUTCOMES:
Quality of life score (EVA scale) of patient's close relatives | 12 months
  difference in gain observed at six months in the mean quality of life score (EVA scale) between close relations having benefited from the PTE program and those having benefited from usual support.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No